CLINICAL TRIAL: NCT02520791
Title: A Phase I Trial of MEDI-570 in Patients With Relapsed/Refractory Peripheral T-Cell Lymphoma (PTCL) Follicular Variant and Angioimmunoblastic T-Cell Lymphoma (AITL)
Brief Title: Anti-ICOS Monoclonal Antibody MEDI-570 in Treating Patients With Relapsed or Refractory Peripheral T-cell Lymphoma Follicular Variant or Angioimmunoblastic T-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01271; NCI-2015-01271 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PJC-021; 9930 (Other: University Health Network Princess Margaret Cancer Center LAO); 9930 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2015-08-10; First posted 2015-08-13 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Advanced Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Recurrent Follicular Helper T-Cell Lymphoma, Angioimmunoblastic-Type; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3a Follicular Lymphoma; Recurrent Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Recurrent Mycosis Fungoides; Recurrent Primary Cutaneous T-Cell Non-Hodgkin Lymphoma; Refractory Follicular Helper T-Cell Lymphoma, Angioimmunoblastic-Type; Refractory Grade 1 Follicular Lymphoma; Refractory Grade 2 Follicular Lymphoma; Refractory Grade 3a Follicular Lymphoma; Refractory Mature T-Cell and NK-Cell Non-Hodgkin Lymphoma; Stage IB Mycosis Fungoides AJCC v7; Stage II Mycosis Fungoides AJCC v7; Stage III Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage III Mycosis Fungoides AJCC v7; Stage IV Cutaneous T-Cell Non-Hodgkin Lymphoma; Stage IV Mycosis Fungoides AJCC v7
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, T-Cell; Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — MEDI-570

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (MEDI-570) (Experimental): Patients receive anti-ICOS monoclonal antibody MEDI-570 IV over 1-4 hours on day 1. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-ICOS Monoclonal Antibody MEDI-570; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Biological: Anti-ICOS Monoclonal Antibody MEDI-570 — Given IV
  Other Names: MEDI-570
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and best dose of anti-inducible T-cell co-stimulator (ICOS) monoclonal antibody MEDI-570 in treating patients with peripheral T-cell lymphoma follicular variant or angioimmunoblastic T-cell lymphoma that has returned after a period of improvement (relapsed) or has not responded to previous treatment (refractory). Immunotherapy with monoclonal antibodies, such as anti-ICOS monoclonal antibody MEDI-570, may induce changes in the body's immune system and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, maximum tolerated dose and recommended phase II dose (RP2D) of anti-ICOS monoclonal antibody MEDI-570 (MEDI-570) in patients with refractory/relapsed peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS), angioimmunoblastic T-cell lymphoma (AITL), follicular lymphoma, mycosis fungoides (MF) and cutaneous T-cell lymphomas (CTCL).

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetic profile of MEDI-570. II. To evaluate the overall response rate (ORR) and progression free survival (PFS) of MEDI-570 at all dose levels and in a 10-patient expansion cohort at the maximum tolerated dose (MTD).

III. To determine short and long term effects of MEDI-570 at all dose levels on the immune system and on T-cell lymphocyte subsets.

IV. To determine the relationship between ICOS expression on tumor cells and response to MEDI-570.

EXPLORATORY OBJECTIVE:

I. To evaluate biomarkers of response and resistance to MEDI-570 in the study population.

OUTLINE: This is a dose-escalation study.

Patients receive anti-ICOS monoclonal antibody MEDI-570 intravenously (IV) over 1-4 hours on day 1. Treatment repeats every 21 days for up to 8 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 weeks for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of one of the following:

  * For dose escalation:

    * Confirmed diagnosis of peripheral T-cell lymphoma (PTCL) or angioimmunoblastic T-cell lymphoma (AITL) that is refractory to at least one line of therapy; anaplastic large cell lymphoma (ALCL) and natural killer T-cell lymphoma nasal type (NKTCL) are excluded
    * Advanced stage cutaneous T-cell lymphoma (CTCL), specifically CTCL NOS, small/medium T-cell lymphoma (SMTCL) and mycosis fungoides (MF) stage IB, IIA, IIB, III and IV that have relapsed after at least one specific prior therapy (e.g. interferon, photopheresis, denileukin difitox, bexarotene, etc); anaplastic cutaneous large cell lymphoma (ACLCL) and lymphomatoid papulopsis are excluded
    * Follicular lymphoma grade 1, 2 or 3A that meets the following criteria:

      * Relapsed or refractory to at least 2 lines of therapy AND
      * Relapsed or refractory post autologous cell transplantation (HCT)
  * For dose expansion/dose confirmation phase:

    * Patients with confirmed diagnosis of peripheral T-cell lymphoma (PTCL) follicular type or angioimmunoblastic T-cell lymphoma (AITL) that is refractory to at least one line of therapy
* At least 14 days from the last therapy dose or 5 half-lives (whichever is shorter), and resolution of toxicity related to the last therapy, excluding grade 2 or less peripheral neuropathy and alopecia; for radiation therapy, a minimum of 2 weeks and resolution of all acute toxicity will be required
* Patients must have at least one measurable lesion that can be accurately measured with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI) scan, or physical exam (by calipers only); (PTCL, AITL and follicular lymphoma patients will be assessed on this study using the Lugano criteria for the evaluation of lymphomas; CTCL and MF patients will be assessed using International Society for Cutaneous Lymphomas [ISCL] and European Organization for Research and Treatment of Cancer [EORTC] criteria)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 6 months
* Leukocytes >= 3,000/mcL
* Hemoglobin >= 80 d/L (or >= 8 g/dL)

  * Patients must not have received a transfusion, with packed red blood cells, within 2 weeks prior to sample being collected
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets (PLT) >= 50,000/mcL
* Absolute CD4 count > 100 cells/uL
* Total bilirubin < 1.5 upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine < 1.5 mg/dl (= 132 umol/L) or
* Creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* In patients with bone marrow involvement the minimum requirement is as follows:

  * Leukocytes >= 2000/mcL
  * ANC >= 1000/mcL
  * PLT >= 50 000/mcL
* Availability of tissue for correlative studies; patients must have at least 6-8 unstained slides of archived formalin-fixed, paraffin-embedded tumor tissue available; if not enough archived tissue is available, a fresh tumor biopsy prior to study initiation is mandatory; for patients who have undergone a fresh baseline biopsy at baseline, the archived tissue is not mandatory
* The effects of MEDI-570 on the developing human fetus are unknown; for this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, during the study participation, and for 3 months after the last dose of the drug; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must have either had a prior vasectomy or agree to use effective contraception prior to the study, during the study, and for 3 months after the last dose of the drug; males should avoid fathering children during and for at least three months after therapy is completed
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who are receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MEDI-570 or history of anaphylaxis to any biological component
* Any history or evidence of opportunistic infection within 6 months of screening including tuberculosis, severe cytomegalovirus (CMV) or herpetic infections (such as disseminated herpes, herpes encephalitis, ophthalmic herpes)
* Evidence of active infection by hepatitis B and/or C; active viral infection by hepatitis B and hepatitis C could be associated with cytopenias (due to hypersplenism or due to the active virus itself), which could add further risk when a potential immunosuppressive medication is used; for patients with hepatitis B treated with anti-virals to undetectable viral load, and for patients with hepatitis C with undetectable ribonucleic acid (RNA) levels and no evidence of liver damage, enrollment may be considered and should discuss first with study's principal investigator
* History of human immunodeficiency virus (HIV) infection; the human immunodeficiency virus (HIV) depletes CD4 T-cells and could also have a role in T-cell anergy; since MEDI-570 preferentially affects CD4 T-cell numbers and function, and the resultant immunosuppression by this agent can be prolonged, exposing HIV patients to MEDI-570 will place them in an unnecessary risk of developing infections due to an underlying acquired cellular immunity defect
* History of primary immunodeficiency
* Receipt of live or live attenuated vaccine within 12 weeks prior to enrollment
* All potential patients must undergo a tuberculosis (TB) test prior to study entry to rule out active or latent tuberculosis (either purified protein derivative [PPD] or QuantiFERON-TB Gold, whichever is preferred and available at the institution); patients with a history of TB (even if treated), or evidence of active or latent TB, are excluded; the diagnosis of active TB is defined per current guidelines; patients with a positive TB test (e.g. PPD or QuantiFERON-TB Gold) will be excluded; patients with history of Bacille-Calmette-Guerin (BCG) vaccination will be tested with QuantiFERON-TB Gold test in order to rule out exposure to TB
* Patients who have undergone allogeneic stem cell transplantation
* Patients who have undergone autologous stem cell transplantation within 3 months from study entry
* Major surgery within 30 days prior or during the study period
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study due to the potential toxicity in pre-clinical reproductive studies; in addition, there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with MEDI-570; breastfeeding should be discontinued if the mother is treated with MEDI-570
* Patients with active, known, or suspected autoimmune disease, except in these conditions:

  * Participants with well-controlled asthma and/or mild allergic rhinitis (seasonal allergies) are eligible
  * Participants with the following disease conditions are also eligible:

    * Vitiligo,
    * Type 1 diabetes mellitus
    * Residual hypothyroidism due to autoimmune condition only requiring hormone replacement
    * Euthyroid participants with a history of Grave's disease (participants suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study drug)
    * For patients with ITP (idiopathic thrombocytopenic purpura) or AIHA (autoimmune hemolytic anemia), a case by case discussion with study principal investigator (PI) may be considered
    * Patients not receiving systemic therapy (i.e., systemic steroids or biologic therapy with disease modifying anti-rheumatic drugs [DMARDs]) within 2 years can be also eligible
* Patients with a weight of < 39 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-09-13 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Incidence of toxicity and safety of anti-inducible T-cell co-stimulator (ICOS) monoclonal antibody MEDI-570 | Up to 12 weeks after completion of study treatment
  Graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest. Adverse events will be summarized using all adverse events experienced, although a sub-analysis may be conducted including only those adverse events in which the treating physician deems possibly, probably or definitely attributable to one or both study treatments.
Maximum tolerated dose (MTD) of anti-inducible T-cell co-stimulator (ICOS) monoclonal antibody MEDI-570 | Up to 21 days
  Toxicity will be assessed using the NCI CTCAE, version 5.0.
Recommended phase 2 dose of anti-inducible T-cell co-stimulator (ICOS) monoclonal antibody MEDI-570 | Up to 21 days
  Toxicity will be assessed using the NCI CTCAE, version 5.0.

SECONDARY OUTCOMES:
Pharmacokinetics (PK), such as plasma concentration and PK parameters, of monoclonal antibody therapy | Prior to dose on day 1, immediately after dose, and at 6 minutes, 24, 48 and 72 hours post dose of cycle 1 and cycle 2, and then on day 1 pre-dose of every subsequent cycle
  Attempts to model associations between pharmacokinetic data with toxicity profiles will be performed primarily using descriptive statistics; however, logistic regression may be used if warranted.
Overall response rate | Up to 36 weeks
  Assessed per the Revised Response Criteria for Malignant Lymphoma of the Lugano Classification. Summary statistics, such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. For all statistical tests, two-sided tests will be performed and no p-value adjustment performed due to the exploratory nature of these tests. A p-value of 0.05 or less will be considered statistically significant.
Progression-free survival | Up to 12 weeks after completion of study treatment
  Summary statistics, such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. For all statistical tests, two-sided tests will be performed and no p-value adjustment performed due to the exploratory nature of these tests. A p-value of 0.05 or less will be considered statistically significant.
Immunogenicity | Up to 36 weeks
  Summary statistics, such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. For all statistical tests, two-sided tests will be performed and no p-value adjustment performed due to the exploratory nature of these tests. A p-value of 0.05 or less will be considered statistically significant.
Overall survival (OS) | Up to 12 weeks after completion of study treatment
  Summary statistics, such as the mean, median, counts and proportion, will be used to describe patients' clinical characteristics. For all statistical tests, two-sided tests will be performed and no p-value adjustment performed due to the exploratory nature of these tests. A p-value of 0.05 or less will be considered statistically significant.

OTHER OUTCOMES:
Biomarkers of response and resistance to anti-inducible T-cell co-stimulator (ICOS) monoclonal antibody MEDI-570 | Up to 36 weeks
  Predictors of clinical outcomes will be investigated using logistic regression, Cox proportional hazards regression and/or generalized estimating equations as appropriate. Potential predictors include clinical predictors and molecular correlates. Descriptive statistics and plotting of data will also be used to better understand potential relationships.

CONTACTS AND LOCATIONS:
Overall Officials: Julio C Chavez, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (23):
- United States (21):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
- Canada (2):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Chavez JC, Foss FM, William BM, Brammer JE, Smith SM, Prica A, Zain JM, Tuscano JM, Shah H, Mehta-Shah N, Geethakumari PR, Wang BX, Zantinge S, Wang L, Zhang L, Boutrin A, Zhao W, Cheng L, Standifer N, Hewitt L, Enowtambong E, Shao W, Sharma S, Carlesso G, Moscow JA, Siu LL. Targeting the Inducible T-cell Costimulator (ICOS) in Patients with Relapsed/Refractory T-follicular Helper Phenotype Peripheral T-cell and Angioimmunoblastic T-cell Lymphoma. Clin Cancer Res. 2023 May 15;29(10):1869-1878. doi: 10.1158/1078-0432.CCR-22-2955. PMID 36826995